CLINICAL TRIAL: NCT06171373
Title: Extension for Menopause Sample Collection
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1415
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will provide urine samples from women going through the menopause transition in order to maintain the SPD sample bank.

Symptom information and cycle length will also be recorded to observe how these change through the menopause transition.

DETAILED DESCRIPTION:
This is an extension to a previous sample collection (Protocol-1326) where additional samples will be collected from the women who continue to go through the menopausal transition (i.e. are not post-menopausal).

Three sets of 10 consecutive daily urine samples will be collected at three timepoints (month 0, month 6 and month 12).

Urine samples will be received in the clinical laboratory and aliquoted into 2.25ml amounts and stored at -80˚C until required.

ELIGIBILITY:
Inclusion Criteria:

* Pre- and peri-menopausal volunteers(assigned by STRAW+10 criteria) who completed PROTOCOL-1326

Exclusion Criteria:

* Post-menopausal volunteers (12 months since last menstrual period)
* Use of hormone replacement therapy (HRT)
* Use of hormone contraception
* Hysterectomy and/or oophorectomy
* Pregnant or breast feeding
* Other medical reason for amenorrhea (absence of menstruation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Study Population: Healthy female volunteers
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Number of Urine Samples Collected | Daily samples for 10 days at 0, 6 and 12 months
  Daily Urine Samples

SECONDARY OUTCOMES:
Menopause Symptom Questionnaire | Recorded at 0, 6 and 12 months
  Experience of a range of menopause symptoms on a 5-point scale (where 1 is very mild and 5 is very severe)

CONTACTS AND LOCATIONS:
Overall Officials: Raniero Zazzeroni, Study Director — SPD Development Company; Jackie Boxer, Principal Investigator — SPD Development Company
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No